CLINICAL TRIAL: NCT04691297
Title: A Digitally-enhanced Smoking Cessation Intervention for High-risk Smokers: Phase II
Brief Title: Digitally Enhanced Smoking Cessation for High Risk Smokers
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: American Association for Cancer Research (Other)
Responsible Party: Principal Investigator, Mary E. Cooley, Phd, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20-457
Record Dates: First submitted 2020-12-17; First posted 2020-12-31 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Smoking; Smoking Cessation; Lung Cancer Screening; Smoking, Tobacco; Smoking Behaviors
Keywords: Smoking; Smoking Cessation; Lung Cancer Screening; Smoking, Tobacco; Smoking Behaviors
MeSH Terms: conditions — Smoking; Smoking Cessation; Tobacco Smoking | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Escape (Experimental): The ESCAPE program provides 8 counseling sessions over the phone, provides nicotine replacement therapy at no cost, and education about lung screening
  Interventions: Other: Escape
- Standard Care (Experimental): The usual care program will include 1 counseling session, nicotine replacement therapy at no cost referral and enrollment in quitworks and an educational brochure about lung cancer screening
  Interventions: Other: Standard Care

INTERVENTIONS:
Other: Escape — The ESCAPE intervention consists of five components:1) behavioral counseling, 2) the use of NRT, 3) digital SNC 4) decision aid about LDCT screening, and 5) a letter and educational materials sent to the primary care provider.
  Arms: Escape
Other: Standard Care — Participants in the standard care arm (brief advice and referral to quit line), will be referred to the MA Quitline which provides free NRT by the study team and will receive an educational brochure related to lung cancer screening.
  Arms: Standard Care

SUMMARY:
This is a research study, is testing a program to improve lung health through smoking cessation and providing education around lung screening.

In this research study involves Studying the Enhanced Smoking Cessation Approaches to Promote Empowerment (ESCAPE) program compared to usual care.

The ESCAPE program was developed help women with HIV quit smoking. Women in the ESCAPE program quit smoking and stayed quit for longer (up to 3 months). For this study, investigators have added a lung screening to the ESCAPE program and want to test if this will improve lung health through increasing quit rates and lung screening.

.

DETAILED DESCRIPTION:
* This is a research study, is testing a program to improve lung health through smoking cessation and providing education around lung screening. The research study procedures include: screening for eligibility and study interventions including participation in counseling and completion of questionnaires by e-mail, phone or in-person.
* This research study involves participating in either the Enhanced Smoking Cessation Approaches to Promote Empowerment (ESCAPE) program or the usual care. Participants will be randomized into one of two groups:

  * ESCAPE: The ESCAPE program provides 8 counseling sessions over the phone, provides nicotine replacement therapy at no cost, and education about lung screening
  * Usual Care: The usual care program will include 1 counseling session, nicotine replacement therapy at no cost referral and enrollment in quitworks
* Participants will be in this research study for up to 6-months.
* It is expected that about 250 people will take part in this research study.

ELIGIBILITY:
Inclusion Criteria:

* 55 to 77 years of age
* No previous history of lung cancer
* ECOG performance status < 2
* ≥ 30 pack year smoking history
* Smoke ≥ 5 cigarettes/day
* Own a mobile phone with access to a video call application
* Has a primary care provider (PCP)
* Provide contact information for the PCP
* Active health insurance
* Has not had LDCT screening
* English speaking
* Can complete an interview

Exclusion Criteria:

* Hospitalization for severe mental illness within the last year.
* The following special populations will not be included

  * Adults unable to consent
  * Individuals who are not yet adults (infants, children, teenagers)
  * Pregnant women
  * Prisoners

Ages: 55 Years to 77 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
7-day point prevalence smoking cessation rate | 3 months
  biochemical verification of smoking status will be done and the %7-day point prevalence abstinence will be compared between two groups with exact binomial test,
7-day point prevalence smoking cessation rate | 6 months
  biochemical verification of smoking status will be done and the %7-day point prevalence abstinence will be compared between two groups with exact binomial test,
number of cigarettes smoked/day | 3 months
  self-report number of cigarettes will be compared with exact Poisson test.
number of cigarettes smoked/day | 6 months
  self-report number of cigarettes will be compared with exact Poisson test.
Lung cancer screening behavior measure | 3 Months
  (stage of low-dose computed tomography [LDCT] screening adoption) Lung Cancer Screening Behaviors[20] will be measured with a questionnaire based on the Precaution Adoption Process Model. This model has seven stages of adoption which includes; stage 1=no awareness of lung cancer screening, stage 2=not engaged with lung cancer screening, stage 3=deciding about action, stage 4= decide not to screen, stage 5=decided to act, stage 6-=acting, and stage 7=maintenance. stage of change will be compared between two groups with exact binomial test,
Lung cancer screening behavior measure | 6 months
  (stage of low-dose computed tomography [LDCT] screening adoption) Lung Cancer Screening Behaviors[20] will be measured with a questionnaire based on the Precaution Adoption Process Model. This model has seven stages of adoption which includes; stage 1=no awareness of lung cancer screening, stage 2=not engaged with lung cancer screening, stage 3=deciding about action, stage 4= decide not to screen, stage 5=decided to act, stage 6-=acting, and stage 7=maintenance. stage of change will be compared between two groups with exact binomial test,

SECONDARY OUTCOMES:
Completion rate | 1 month
  The evaluation of the storytelling narrative communication at 1 and 3 months will be defined as follows:1) > 80% receipt and completion rate of watching the SNC digitalized videos.
  Descriptive statistics (estimate and 95% CI) will be used to report completion rate.
Completion rate | 3 months
  The evaluation of the storytelling narrative communication at 1 and 3 months will be defined as follows:1) > 80% receipt and completion rate of watching the SNC digitalized videos.
  Descriptive statistics (estimate and 95% CI) will be used to report completion rate.
Percentage of the group perceive the film as just right in length | 1 month
  defined as > 80% of the group perceive the film as just right in length in addition to favorable comments, the Narrative Engagement Scale scores are ≥ to the established means ). Descriptive statistics (estimate and 95% CI) will be used to report percentage and one-sample t-test will be used to compare Narrative Engagement Scale scores to the established means.
Percentage of the group indicate that the film would have value to others | 3 months
  > 80% of the group comments indicate that the film would have value to others and the Narrative Engagement Scale scores are ≥ to the established means. Descriptive statistics (estimate and 95% CI) will be used to report percentage and one-sample t-test will be used to compare Narrative Engagement Scale scores to the established means.
Narrative Engagement Scale scores | 1 month
  The ratings of SNC videos will be evaluated using the Narrative Engagement Scale that will be administered at 1 and 3 months [37] The scale is a paper and pencil questionnaire developed to measure the extent to which the viewer of narratives in a variety of forms (film, TV etc.) becomes engaged, transported, or immersed in the narrative and the potential of the narrative to affect change in story-related attitudes and beliefs. The scale scores range from 1-7 with 7 indicating greater engagement.
Narrative Engagement Scale scores | 3 months
  The ratings of SNC videos will be evaluated using the Narrative Engagement Scale that will be administered at 1 and 3 months [37] The scale is a paper and pencil questionnaire developed to measure the extent to which the viewer of narratives in a variety of forms (film, TV etc.) becomes engaged, transported, or immersed in the narrative and the potential of the narrative to affect change in story-related attitudes and beliefs. The scale scores range from 1-7 with higher scores indicating greater engagement.
Polygenic risk score (PRS) | 6 months
  We will construct three PRS. The first will be based on the lead single nucleotide polymorphisms (SNPs) from 183 independent genetic loci associated at genome-wide significance (p<5x10-8) with ever smoking status in adults from the UK Biobank and the Tobacco and Alcohol Genetic Consortium. The risk will be calculated as the weighted sum of each genetic variant, under an additive genetic model, counting the number of copies of the risk increasing allele. The weights will be proportional to the estimated effect size of each SNP. The second risk score will be constructed from a larger set of SNPs (~1 million) from the same GWAS using LDPred that allows for the construction of more powerful PRSs for specific racial groups using linkage disequilibrium information from large genetic reference panels. Finally, we will also construct a PRS based on the GWAS results for the largest available study specifically for nicotine dependence using the LDPred approach.
Qualitative interviews | 6 months
  A semi-structured interview will be conducted with participants. Topics for the interview guide include; 1) perceptions of genomic evaluation, 2) experiences for providing risk information, 3) preferences for receiving risk information, 4) experiences with the study interventions, 5) suggestions for program improvements.

CONTACTS AND LOCATIONS:
Overall Officials: Mary E. Cooley, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu